CLINICAL TRIAL: NCT00503945
Title: The Clinical Significance of an Index of Cardiac Function, Tei-Index, in Obstructive Sleep Apnea Syndrome Patients.
Brief Title: Cardiac Dysfunction in Obstructive Sleep Apnea Patients: Prevalence of and Effect of nCPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nagasaki University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nagasaki-SAS
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2007-07-19 (Estimated); Status verified 2007-07

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; continuous positive airway pressure; echocardiography; Natriuretic peptide
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Nasal continuous positive airway pressure (nCPAP)

SUMMARY:
The aim of this study is to clarify the influence of obstructive sleep apnea syndrome on left ventricular function using echocardiographic parameters including the myocardial performance index (Tei-index), and to determine the short-term effects of nCPAP on them.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) affects 2% and 4% of middle-aged women and men respectively, and is associated with an increased risk of cardiovascular complications. Therefore, cardiovascular consequences must be evaluated in the clinical management of OSAS and the study of cardiac functional parameters could be particularly useful. Reported findings are conflicting with respect to the influence of OSAS and nasal continuous positive airway pressure (nCPAP) on left ventricular function. In this study, we assess cardiac dysfunction with echocardiographic parameters, such as LVEF, left ventricular mass, ratio of E to A (E/A) and mitral deceleration time (DT) from the mitral inflow velocity, and Tei-index, or plasma brain natriuretic peptide (BNP) level at baseline, and 1 and 3 months after nCPAP treatment. The main endpoint is the comparison of echocardiographic parameters and BNP between OSAS patients and control subjects, and the changes of them after short-term of nCPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* OSAS patients: Moderate to severe OSAS patients with apnea-hypopnea index (AHI) ≥ 20 events/hour by overnight polysomnography and start nCPAP treatment.

Exclusion Criteria:

* Apparent lung diseases
* Daytime hypoxemia (PaO2 <80 mmHg)
* Atrial fibrillation, bundle branch block, atrioventricular block and implantable pacemaker
* Left ventricular dysfunction (ejection fraction <50%)
* Ischemic or valvular heart disease, and cardiomyopathy determined from medical history or a physical examination, electrocardiogram (ECG), chest radiography, and echocardiography
* Renal insufficiency (serum creatinine >2.0 mg/dl).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-11; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Effect of nCPAP treatment on echocardiographic parameters including LVEF, left ventricular mass, ratio of E to A (E/A) and mitral deceleration time (DT) from the mitral inflow velocity, and Tei-index. | baseline, 1 month, 3months

SECONDARY OUTCOMES:
Effect of nCPAP treatment on plasma brain natriuretic peptide (BNP) level. | baseline, 1 month, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Ikeda, M.D., Ph.D., Study Chair — Second Department of Internal Medicine, Nagasaki University School of Medicine
Locations (1):
- Second Department of Internal Medicine, Nagasaki University School of Medicine, Nagasaki, Japan